CLINICAL TRIAL: NCT05909033
Title: Early Predictors for the Short Term Native Liver Survival in Patients With Biliary Atresia After Kasai Procedure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weibing Tang (Other)
Responsible Party: Sponsor-Investigator, Weibing Tang, Clinical Professor, Nanjing Children's Hospital
Organization: Nanjing Children's Hospital (Other)
Other Study IDs: NanjingCH20230601
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Biliary Atresia
Keywords: biliary Atresia; Kasai procedure; early predictor; native liver survival
MeSH Terms: conditions — Biliary Atresia | interventions — Portoenterostomy, Hepatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Kasai procedure — All KPs were performed by a medical team. This technique involved creation of a 35-40 cm Roux loop to facilitate biliary drainage. After dissection of the hepatic vasculature at the hilum and excision of the hilar plate, hepaticojejunostomy was performed as an anastomosis extending from the bifurcation of the right hepatic artery into anterior and posterior branches to the Rex confluence of the left portal vein with the obliterated umbilical vein.

SUMMARY:
Many factors have been proven that may affect NLS in BA patients after KP;however,the early predictors for NLS were not be finally detected.This study was designed to evaluate and identify the preoperative and early postoperative factors associated with NLS for early prediction in BA patients after KP.

DETAILED DESCRIPTION:
Biliary atresia (BA) is the most common cause of neonatal cholestasis, occurring in approximately 1: 8000 to 1:15000 in Asian populations compared with those in Europe and the USA, with a ratio of 1: 1.56 in males and females.Until now, Kasai procedure(KP) remains the preferred treatment for biliary BA;however,nearly 60-70% patients after KP need liver transplants to achieve long-term survival.Therefore, it is meaningful to seek and analyze the factors affecting the native liver survival(NLS) in BA patients with KP for prediction. Luckily， A lot of studies have designed to seek the risk factors for death or liver transplants in BA patients after KP,and many factors have been proven that may affect NLS,including old age at KP,low gamma-glutamyl transpeptidase(GGT) level,Cytomegalovirus(CMV) Infection,early jaundice clearance(JC) and postoperative cholangitis(PC),etal.However,the predictors for NLS were not be finally detected.Otherwise,the safety of liver transplants has been improved in the past few years and performing liver transplant in young infants has been proven to be feasible.Then,it is important to seek early NLS predictors for counseling the necessity and timing of liver transplant.Unfortunately,early predictors of NLS focus on preoperative and early postoperative period after KP were insufficient.

This study is primarily designed to evaluate and identify the preoperative and early postoperative factors associated with NLS for early prediction in BA patients after KP.

ELIGIBILITY:
Inclusion Criteria:

Biliary Atresia(BA) patients performed with Kasai Procedure patients completed the follow-up>6 months

Exclusion Criteria:

BA patients without KP patients lost of follow-up BA patients with other severe complications lead to death

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with Biliary atreisa and were performed with kasai procedures
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
NLS rate | through study completion, an average of 3 years
  native liver survival rate

SECONDARY OUTCOMES:
age at KP | through study completion, an average of 3 years
  age at kasai procedure
PC | through study completion, an average of 3 years
  post cholangitis
JC | through study completion, an average of 3 years
  jaudiance clearance

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Tang, Dr, Study Director — Children's Hospital of Nanjing Medical University; Weibing Tang, Dr, Principal Investigator — Children's Hospital of Nanjing Medical University
Locations (1):
- Children's Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Lu C, Xie H, Zhu Z, Ding Z, Geng Q, Tang W. A convenient nomogram for predicting early death or liver transplantation after the Kasai procedure in patients with biliary atresia. Langenbecks Arch Surg. 2024 Jan 8;409(1):30. doi: 10.1007/s00423-023-03216-5. PMID 38189999